CLINICAL TRIAL: NCT03770598
Title: Team Based Psychosocial Care to Promote, Maintain and Restore Wellness of Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Shehzad K. Niazi, Prinicpal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-000718
Record Dates: First submitted 2018-11-19; First posted 2018-12-10 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
Keywords: Psychosocial Care; Wellness
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Non-Distressed patients will be randomized to receive intervention or standard of care.
  Distressed patients will be randomized to receive intervention or standard of care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Distressed (Active Comparator): Study participants who do indicate distress or who do meet criteria for depression or anxiety will be randomized to receive either treatment as usual (referral to Psychiatry or Psychology for evaluation and further treatment) or team based care model.
  Interventions: Behavioral: Standard of Care Distressed in study Arm Distressed; Behavioral: Team Based Care
- Non-Distressed (Active Comparator): Study participants who do not indicate distress or who do not meet criteria for depression or anxiety will be randomize to monitoring only or to receive psycho-education regarding subjects that when used can promote wellness.
  Interventions: Behavioral: Psycho-Education; Behavioral: Standard of Care Non-Distressed

INTERVENTIONS:
Behavioral: Standard of Care Distressed in study Arm Distressed — Social worker evaluation and possible referral to Psychiatry/Psychology for evaluation and further treatment.
  Arms: Distressed
Behavioral: Psycho-Education — Mindfulness based stress reduction class, yoga and education material
  Arms: Non-Distressed
Behavioral: Team Based Care — Psychiatrist, Oncologist, clinical social worker, study coordinator
  Arms: Distressed
Behavioral: Standard of Care Non-Distressed — No psycho-education about wellness promotion or health. These patients will be monitored only.
  Arms: Non-Distressed

SUMMARY:
Researchers are trying to see if proactive identification and team based individualized care of cancer patients having emotional difficulties can improve quality of life relative to treatment as usual. Also, to see if proactive approaches to maintain wellness can prevent grief among breast cancer patients, experiencing no emotional difficulties relative to treatment as usual.

DETAILED DESCRIPTION:
Consented subjects will be randomized into two separate groups. Groups will be distressed and non-distressed subjects. Each group will be randomized into either intervention education training or standard of care. Both groups will be asked to fill out questionnaires during the duration of the study. Subjects will be remain in the study for up to one year.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of breast cancer within last three years
* Able to communicate in English or with the help of an interpreter.
* Access to a device with internet connection

Exclusion Criteria:

* Breast cancer patients who are considered for hospice or expected survival of less than six months.
* Presence of active suicidal ideations.
* Presence of active psychosis.
* Presence of dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2021-11-16 (Actual); Study Completion 2021-11-16 (Actual)

PRIMARY OUTCOMES:
Change in Wellness | baseline, 6 months
  Subject wellness scores based on Short Warwick-Edinburgh Mental-Wellbeing Scale. This is a 7 item scale monitoring of mental wellbeing in subjects. Responses are based on a 1 to 5 item scale with 1 = None of the time, 2 = Rarely, 3 = Some of the Time, 4 = Often, 5 = All of the Time.

SECONDARY OUTCOMES:
Improvement in depression compared to baseline | one year
  measured by using PHQ-8 (Patient Health Questionnaire); this is an 8 item scale. Scores of 5 or less are considered no depression, 5-10, mild depression, 11-15, moderate depression, 16-20 moderately severe and more than 20 is considered severe depression.
Improvement in anxiety compared to baseline | One Year
  Will be measured by GAD-7 (Generalized Anxiety Disorder 7-item Scale). Its a 7 item scale. Cut points of 5, 10, 15 represent mild, moderate and severe levels of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Shehzad K Niazi, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials